CLINICAL TRIAL: NCT03808142
Title: PROmyBETAappGame: Ascertaining Medication Usage & Patient Reported Outcomes Via the myBETAapp and Exploring Gamification in Patients With Multiple Sclerosis Treated With Betaferon
Brief Title: PROmyBETAappGame: a Study to Learn More About the Medication Usage & Patient Reported Outcomes Via the myBETAapp and to Find Out More About the Usage of Game Principles and Game Design Elements (Gamification) in Medical Care of Patients With Multiple Sclerosis Treated With Betaferon
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20263
Record Dates: First submitted 2019-01-10; First posted 2019-01-17 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: During a 3-months period all patients with an active myBETAapp account were invited to participate in the study (3-month invitation period=enrollment period). Patients seek more information about the study were able to access a detailed informed consent form via their app providing step-by-step background information. Those patients were wishing to participate in the study were able to provide (electronic) informed consent (ICF).
  Interventions: Other: myBETAapp; Other: PEAK; Drug: Betaferon, BAY86-5046; Device: BETACONNECT

INTERVENTIONS:
Other: myBETAapp — Patients choosing to use the myBETAapp were required to insert the Mixject number from their prescribed Betaferon box, which serves as an opening key for the app. Obtaining a new Betaferon box and obtaining a new Mixject number was not interfere with the process of continuously allocating data to a single patient; each patient had a unique personal identifier in the database. All data recorded in the myBETAapp including demographic and injection-related data were stored in the database once the mobile device was connected to the internet.
Other: PEAK — Peak is an application that aims at helping its users to challenge their brains and keep them sharp.
Drug: Betaferon, BAY86-5046 — Injection
Device: BETACONNECT — BETACONNECT automatically records and stores injection-related details including injection time, speed, and depth upon every injection.

SUMMARY:
In this study researchers wanted to learn more about the medication usage behavior among multiple sclerosis (MS) patients treated with Betaferon using the myBETAapp which includes the elements to what extent

* taking medication matched the presciber´s recommendation (adherence, compliance),
* treatment for the prescribed duration (persistence) was continued and
* injections were missed. Among MS patients treated with Betaferon using the myBETAapp the study also collected information on the health-related quality of life, treatment satisfaction and satisfaction with treatment support.

DETAILED DESCRIPTION:
The PROmyBETAappGame study was a mixed prospective and retrospective, non-interventional, observational cohort study

ELIGIBILITY:
Inclusion criteria

* Patients aged ≥ 18 years.
* Patients on treatment with Betaferon (every Betaferon box contains a "Mixject" number, which is a product specific number unrelated to the study. Only patients prescribed Betaferon for their MS will be able to use the myBETAapp and participate in the study).
* Patients must be using the myBETAapp.
* Electronic informed consent must be obtained.

Exclusion criteria

- No exclusion criteria for participation in this study were defined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women and men in Germany with the diagnosis of MS that were treated with Betaferon and used the myBETAapp were eligible to participate in the study. The option to enroll in the study was offered after log-in procedure to myBETAapp.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-09-02 (Actual)

PRIMARY OUTCOMES:
Compliance percentage to therapy | Up to 12 months from informed consent provided
  Assessed prospectively
Persistence percentage of therapy | Up to 12 months from informed consent provided
  Assessed prospectively
Adherence percentage to therapy, assessed prospectively | Up to 12 months from informed consent provided
  Assessed prospectively
Absolute number of injections missed per 3-month intervals | Up to 12 months from informed consent provided
  Assessed prospectively
Relative proportion of injections missed per 3-month intervals | Up to 12 months from informed consent provided
  Assessed prospectively

SECONDARY OUTCOMES:
Compliance percentage to therapy | Retrospective analysis from 01-Sep-2015 to 15-Apr-2019
  Assessed retrospectively
Persistence percentage of therapy | Retrospective analysis from 01-Sep-2015 to 15-Apr-2019
  Assessed retrospectively
Adherence percentage to therapy | Retrospective analysis from 01-Sep-2015 to 15-Apr-2019
  Assessed retrospectively
Absolute number of injections missed per 3-month intervals | Retrospective analysis from 01-Sep-2015 to 15-Apr-2019
  Assessed retrospectively
Relative proportion of injections missed per 3-month intervals | Retrospective analysis from 01-Sep-2015 to 15-Apr-2019
  Assessed retrospectively
Health-related quality of life assessed by questionnaire EQ-5D-5L | Up to 12 months from informed consent provided
  Five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
  Each dimension has 5 levels: (1) no problems , (2) slight problems, (3) moderate problems, (4) severe problems and (5) extreme problems.
Scores of Treatment Satisfaction Questionnaire for Medication version 2 (TSQM v.II) | Up to 12 months from informed consent provided
Response level of Satisfaction with the BETAPLUS patient support program (service questionnaire) | Up to 12 months from informed consent provided
  This question can be answered on a 5-point Likert Scale (Very satisfied/satisfied/neither satisfied nor dissatisfied/ dissatisfied/ very dissatisfied) also including the option "not participating".
Response level of Satisfaction with the BETACONNECT autoinjector (service questionnaire) | Up to 12 months from informed consent provided
  This question can be answered on a 5-point Likert Scale (Very satisfied/satisfied/neither satisfied nor dissatisfied/ dissatisfied/ very dissatisfied) also including the option "not using".
Response level of Satisfaction with the myBETAapp (service questionnaire) | Up to 12 months from informed consent provided
  This question can be answered on a 5-point Likert Scale (Very satisfied/satisfied/neither satisfied nor dissatisfied/ dissatisfied/ very dissatisfied).
Feedback based on free text on supporting services or devices | Up to 12 months from informed consent provided
  Single question
Number of MS patients using the mobile-based cognitive training tool - PEAK | Up to 12 months from informed consent provided
Proportion of MS patients using the mobile-based cognitive training tool - PEAK | Up to 12 months from informed consent provided
Frequency of mobile-based cognitive training tool - PEAK usage (trainings/week) | Up to 12 months from informed consent provided
Duration of mobile-based cognitive training tool - PEAK usage (days) | Up to 12 months from informed consent provided
Cumulative time played per game of mobile-based cognitive training tool - PEAK usage (minutes) | Up to 12 months from informed consent provided

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/